CLINICAL TRIAL: NCT06994507
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Phase 3 Trial of GM1 Prophylaxis for Nab-paclitaxel-associated Chemotherapy-induced Peripheral Neuropathy (CIPN) in Patients With Breast Cancer（Gypsophila )
Brief Title: GM1 Prophylaxis for Nab-paclitaxel-associated Chemotherapy-induced Peripheral Neuropathy (CIPN) in Patients With Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QLGM1-CIPN-301
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GM1 400mg (Experimental): Albumin-paclitaxel was administered on Day 1 of each cycle, Q3W. GM1 is administered with D-1,D1,D2 every cycle
  Interventions: Drug: GM1
- Placebo (Placebo Comparator): Albumin-paclitaxel was administered on Day 1 of each cycle, Q3W. Placebo is administered with D-1,D1,D2 every cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GM1 — GM1 was administered intravenously one day before the administration of each cycle of chemotherapy. The experimental group was given 400 mg of GM1 injection. Administration was carried out at D-1, D1, D2 in each cycle, with a cumulative administration of 3 times per cycle.
  Arms: GM1 400mg
Drug: Placebo — Placebo was administered intravenously one day before the administration of each cycle of chemotherapy. The control group was given placebo. Administration was carried out at D-1, D1, D2 in each cycle, with a cumulative administration of 3 times per cycle.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, multicenter, placebo-controlled phase III clinical trial, aiming to evaluate the efficacy and safety of GM1 in preventing chemotherapy-induced peripheral neuropathy in breast cancer patients treated with Albumin-paclitaxel chemotherapy regimen.

DETAILED DESCRIPTION:
This study was randomly divided into two groups at a ratio of 1:1, with 176 subjects in each group. All patients received GM1/ placebo treatment + chemotherapy.

The main purpose of this study is to evaluate the effectiveness of GM1 in preventing peripheral neuropathy caused by albumin-paclitaxel chemotherapy. The primary endpoint was the end of GM1 treatment in cycle 4 (C4D21), and the proportion of patients whose FACT/GOG-Ntx score changed by more than 12 points from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form;
* Age: 18 to 75 years old;
* Female patients with breast cancer confirmed byhistological and/or cytological diagnostic basis for breast cancer and are intended to receive adjuvant/neoadjuvant therapy with Albumin paclitaxel regimens;
* ECOG: 0-1
* Adequate organ function level
* Glycated hemoglobin (HbA1c) < 7.0%;
* For women of childbearing potential: use effective contraceptive measures for contraception from the date of signing the informed consent form until 30 days after the last use of the investigatory drug.
* Patients can accurately record or express the occurrence and severity of peripheral neuropathy through questionnaires.

Exclusion Criteria:

* Grade ≥1 peripheral neuropathy (CTCAE grade ≥1) or any of the first 4 items of FACT/GOG-Ntx ≥1;
* There are risk factors for peripheral neuropathy (excluding peripheral neuropathy caused by chemotherapy).
* History of another malignant tumors (except breast cancer)
* Symptoms such as muscle pain in the limbs that interfere with the evaluate of peripheral neuropathy;
* Uncontrolled cardiovascular and cerebrovascular system diseases or hypertension
* Active infections that require systematic treatment, including bacteria, fungi or viruses, within one week before first study drug use; Or infectious diarrhea occurred within 4 weeks before the first study drug use;
* Hereditary abnormal glycolipid metabolism, HIV infection or known Acquired Immune Deficiency Syndrome (AIDS); Positive syphilis antibody, active hepatitis B, active hepatitis C

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
FACT/GOG-Ntx scores with a change of more than 12 points from the baseline | At the end of Cycle 4 (21day/Cycle）
  The proportion of those whose FACT/GOG-Ntx score changed by more than 12 points from the baseline at the end of the fourth cycle of treatment

SECONDARY OUTCOMES:
The incidence of grade ≥2 (CTCAE) CIPN | At the end of Cycle 4 (21day/Cycle）,At the end of Cycle 6 (21day/Cycle）
  The incidence of grade ≥2 (CTCAE) CIPN
Assessment of functional impairment | At the end of Cycle 4 (21day/Cycle）,At the end of Cycle 6 (21day/Cycle）
  Vibration sensitivity test and Grooved pegboard test
Assessment of Quality of Life | At the end of Cycle 4 (21day/Cycle）,At the end of Cycle 6 (21day/Cycle）
  Assessment of Quality of Life（QLQ C30）
FACT/GOG-Ntx scores with a change of more than 12 points from the baseline | At the end of Cycle 6 (21day/Cycle）
  The proportion of those whose FACT/GOG-Ntx score changed by more than 12 points from the baseline at the end of the sixth cycle of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of the Chinese People's Liberation Army General Hospital, Beijing, China